CLINICAL TRIAL: NCT02152475
Title: PDT With Blue Light and Curcumin for Oral Disinfection
Brief Title: Photodynamic Therapy (PDT) for Oral Disinfection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Fernanda Rossi Paolillo, Ph.D, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNPQ2013
Record Dates: First submitted 2014-05-24; First posted 2014-06-02 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
Keywords: Blue-LED; Curcumin; PDT; Oral disinfection
MeSH Terms: interventions — Mouthwashes; Curcumin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PDT with blue light and curcumin (Experimental): PDT treatment was performed with light and curcumin.The irradiation parameters were: blue-light emitting diode (LED) illumination (455±30 nm), 400 mW of average optical power, 5 min of application, illumination area of 0.666 cm2, 600 mW/cm2 of intensity and 120 J/cm2 of fluence. The curcumin concentration of 30 mg/L was used.
  Interventions: Drug: mouthwash with curcumin; Device: blue LED illumination
- Curcumin (Active Comparator): The curcumin concentration of 30 mg/L was used.
  Interventions: Drug: mouthwash with curcumin
- Blue light (Active Comparator): The irradiation parameters were: blue-light emitting diode (LED) illumination (455±30 nm), 400 mW of average optical power, 5 min of application, illumination area of 0.666 cm2, 600 mW/cm2 of intensity and 120 J/cm2 of fluence.
  Interventions: Device: blue LED illumination

INTERVENTIONS:
Drug: mouthwash with curcumin — Mouthwash with 20 ml of curcumin solution for 5 minutes
  Arms: Curcumin; PDT with blue light and curcumin
Device: blue LED illumination — Oral cavity was illuminated with blue light for 5 minutes
  Arms: Blue light; PDT with blue light and curcumin

SUMMARY:
Photodynamic therapy (PDT) is a technique used for the oral disinfection. In dentistry, PDT for microbial inactivation may reduces both dental plaque and risk of developing caries as well as contributes to treat gingivitis, periodontitis, peri-implantitis and endodontic diseases. The investigators hypothesis was that PDT with blue light and curcumin promotes oral disinfection during 2 hours after treatment.

DETAILED DESCRIPTION:
PDT uses a non-toxic drug that is activated by exposure to light in the presence of oxygen. The excited state this drug transfers energy or electrons to ground state molecular oxygen producing cytotoxic effects on cell. There are productions of reactive oxygen species (ROS) and disrupts several of the cell's functions. This results in bacterial disinfection. In order to perform the PDT on the oral cavity, a device based on blue LED with transparent acrylic diffuser tip and cylindrical shape was developed.

ELIGIBILITY:
Inclusion Criteria:

* non-users of any antibiotic therapy
* those who do not perform any oral hygiene, such as flossing, brushing and antiseptic mouthwash
* those who performed 12-hour fasting prior the treatment and measurements

Exclusion Criteria:

* oral cancer
* smoking habits
* pregnancy
* patients with partial or total dentures
* orthodontic brackets users

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-05; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Microbiological analysis by the total number of colony-forming units (CFU). | Two hours
  Two saliva samples from each volunteer were collected. The saliva samples underwent serial dilutions and 100-microliters aliquots were plated on brain heart infusion agar plates (in duplicate) and then incubated under microaerophilic conditions. After incubation, the total number of colony-forming units (CFU) was determined.

CONTACTS AND LOCATIONS:
Overall Officials: Vanderlei S Bagnato, Ph.D, Study Director — Physics Institute of São Carlos (IFSC), University of São Paulo (USP); Diego PV Leite, DDS, Principal Investigator — Physics Institute of São Carlos (IFSC), University of São Paulo (USP); Fernanda R Paolillo, Ph.D, Principal Investigator — Physics Institute of São Carlos (IFSC), University of São Paulo (USP); Carla R Fontana, Ph.D, Principal Investigator — Univ Estadual Paulista (UNESP); Thiago Parmesano, Student, Study Chair — Physics Institute of São Carlos (IFSC), University of São Paulo (USP)
Locations (1):
- Fernanda Rossi Paolillo, São Carlos, São Paulo, Brazil

REFERENCES:
- [Result] Araujo NC, Fontana CR, Gerbi ME, Bagnato VS. Overall-mouth disinfection by photodynamic therapy using curcumin. Photomed Laser Surg. 2012 Feb;30(2):96-101. doi: 10.1089/pho.2011.3053. Epub 2012 Jan 6. PMID 22224655
- [Result] Araujo NC, Fontana CR, Bagnato VS, Gerbi ME. Photodynamic antimicrobial therapy of curcumin in biofilms and carious dentine. Lasers Med Sci. 2014 Mar;29(2):629-35. doi: 10.1007/s10103-013-1369-3. Epub 2013 Jun 23. PMID 23793414
- [Result] Gursoy H, Ozcakir-Tomruk C, Tanalp J, Yilmaz S. Photodynamic therapy in dentistry: a literature review. Clin Oral Investig. 2013 May;17(4):1113-25. doi: 10.1007/s00784-012-0845-7. Epub 2012 Sep 27. PMID 23015026
- [Result] Fontana CR, Lerman MA, Patel N, Grecco C, Costa CA, Amiji MM, Bagnato VS, Soukos NS. Safety assessment of oral photodynamic therapy in rats. Lasers Med Sci. 2013 Feb;28(2):479-86. doi: 10.1007/s10103-012-1091-6. Epub 2012 Mar 31. PMID 22467011
- [Result] Soukos NS, Som S, Abernethy AD, Ruggiero K, Dunham J, Lee C, Doukas AG, Goodson JM. Phototargeting oral black-pigmented bacteria. Antimicrob Agents Chemother. 2005 Apr;49(4):1391-6. doi: 10.1128/AAC.49.4.1391-1396.2005. PMID 15793117
- See also: Optics and Photonics Research Center — http://cepof.ifsc.usp.br/